CLINICAL TRIAL: NCT01895114
Title: Assessment of Renal Function in Cirrhotic Patients -A Comparison of Cystatin C and Creatinine Based Calculations to 125I-iothalamate
Brief Title: Assessment of Renal Function in Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 010-263
Record Dates: First submitted 2013-02-11; First posted 2013-07-10 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2015-07

CONDITIONS: Liver Failure; Renal Failure
Keywords: Renal function; cirrhotic patients; transplant evaluation
MeSH Terms: conditions — Liver Failure; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to help determine whether cystatin C is a more sensitive laboratory measurement for renal function in cirrhotic patients.

DETAILED DESCRIPTION:
Serum cystatin C, creatinine clearance based calculations, and 125I-Iothalamate clearance (Glofil) will be obtained in 220 patients with cirrhosis. Utilizing this information, the correlation between cystatin C and 125I-Iothalamate clearance will be obtained. In addition, the current serum creatinine based calculations and true creatinine clearance will also be correlated with 125I-Iothalamate clearance. The results of this study should help to determine whether serum cystatin C is a more sensitive laboratory measurement of renal function in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* over 18 undergoing evaluation for a liver transplant

Exclusion Criteria:

* known allergy or sensitivity to 125I-Iothalamate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Baylor All Saints Medical Center and Baylor University Medical Center who have cirrhosis and a stable urine creatinine
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2010-12; Primary Completion 2021-04 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Creatinine based blood and urine laboratory tests as a measure of renal function in patients with chirrosis of the liver. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fischbach, MD, Principal Investigator — Baylor All Saints
Locations (1):
- Baylor All Saint's Medical Center in Fort Worth, Fort Worth, Texas, United States